CLINICAL TRIAL: NCT03236389
Title: Brain Dynamics in Response to Jugular Vein Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016-6895
Record Dates: First submitted 2017-01-10; First posted 2017-08-01 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Concussion, Mild
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collar Wearing (Experimental): subjects will wear collar during MRI testing
  Interventions: Device: Q Collar

INTERVENTIONS:
Device: Q Collar — measuring changes in brain during MRI while wearing the Q collar

SUMMARY:
Clinical trials have suggested that this device is effective in mitigating changes in brain structure and function in athlete populations. The purpose of the current study is to better understand the underlying mechanistic response of the brain hemodynamics to mild jugular vein compression

DETAILED DESCRIPTION:
Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). A simple, effective, and lightweight device worn by athletes or war fighters in the field, designed to mitigate TBI resulting from blast trauma or concussive events, would save lives, and the huge costs currently being experienced for life-treatment of surviving victims. An externally-worn medical device (the Device) that applies mild jugular vein compression according to the principle of the Queckenstedt Maneuver, is being developed by Q30 Sports Science, LLC (Q30). Preliminary research suggests that the Device has the potential to reduce the likelihood of TBI. The currently developed collar (Smith 2009, Smith and Fisher 2011, Smith and Fisher 2011, Smith 2012) has been approved for studies in humans (IRB 2013-2240) and the results indicate safety for use during high demand and maximal exertion activities. Regarding safety, the externally worn collar is meticulously designed to mimic the body's own omohyoid muscle actions upon the jugular veins that will provide similar pressure and volume increases not to surpass that of a yawn or the mere act of just lying down. Initial safety testing and early clinical trials indicate that the collar application is both safe and efficacious to prevent brain microstructure and neurophysiological changes in response to head impacts.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy volunteer aged 7-40
* Able to provide written consent
* Able to tolerate hypercapnia for 1-2 minutes

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or severe head trauma as indicated through pre-season screening:
* Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Any known airway obstruction
* Any known seizure disorder

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Changes in brain structure while wearing Q collar seen via MRI | immediate
  measure changes in brain structure on MRI

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Cincinnati Childrens Hospital
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No